CLINICAL TRIAL: NCT03328676
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Trial to Investigate the Efficacy and Safety of Avidekel Oil for the Treatment of Subjects With Agitation Related to Dementia
Brief Title: The Effect of Cannabis on Dementia Related Agitation and Aggression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TO Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TO_D02_2016
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Agitation Related to Dementia
MeSH Terms: interventions — nabiximols; Olive Oil; Chlorophyll

STUDY DESIGN:
Intervention Model Description: A Phase II, Randomized, Double-blind, Placebo-controlled Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Avidekel " cannabis oil 20:1 CBD:THC (Experimental): The cannabis oil will be mad out of extract from the Avidekel strain and olive oil. Avidekel oil containing Δ9-Tetra-Hydrocannabinol (Δ9-THC) and Cannabidiol (CBD) in a 1:20 ratio and at a concentration of 30% CBD and 1.5% Δ9-THC. Each Avidekel oil drop is approximately 0.04 ml in volume containing about 12 mg CBD and 0.6 mg Δ9-THC.
  Interventions: Drug: Cannabis
- placebo oil (Placebo Comparator): Patients in the control group will receive placebo.
  Interventions: Drug: Placebo oil

INTERVENTIONS:
Drug: Cannabis — Patients will receive study medication as drops applied under the tongue 3 times a day - morning, noon and evening, at a minimum of 4hr apart between administrations.
  Other Names: CBD-A
  Arms: "Avidekel " cannabis oil 20:1 CBD:THC
Drug: Placebo oil — Patients will receive study medication as drops applied under the tongue 3 times a day - morning, noon and evening, at a minimum of 4hr apart between administrations.
  Other Names: olive oil and chlorophyll
  Arms: placebo oil

SUMMARY:
The most common syndrome in patients with severe dementia is agitated behavior, which is often characterized by a combination of violent behavior (physical or verbal), restlessness, and inappropriate loudness. The treatment options for this syndrome are limited and lead to severe side effects. In vivo experiments on animals and clinical studies on adults show that cannabinoids could have a beneficial effect on behavioral disorders in general, and in dementia-related disorders in particular.

Additionally, medical cannabis patients have reported that cannabis aids in pain relief, increased appetite, and a sense of calm and peace of mind. Elderly patients suffering from dementia that experience this syndrome could also benefit from other quality of life aspects of the cannabis treatment such as reduction in medication consumption, weight gain and improvement of sleep.

DETAILED DESCRIPTION:
In this randomized, double-blind placebo-controlled trial, 60 patients will be randomly assigned to receive either CBD-A (30:1) cannabis rich low THC oil (30% CBD and 1% THC) or a placebo oil. The primary efficacy endpoint was a decrease of four or more points on the Cohen-Mansfield Agitation Inventory (CMAI) score by week 16, as compared to baseline. Secondary endpoints included improvement of other neurobehavioral symptoms.

The following questionnaires will be administered by trained staff at every visit: The CMAI, a to measure the types and frequencies of agitated behaviors, and the Neuropsychiatric Inventory-Nursing Home Version (NPI-NH) to measure behavioral disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > 60 years old.
* Written informed consent from participants legally authorized representative.
* Subjects who are residing either in an institutionalized setting (e.g. dementia unit, nursing home, assisted living facility, or other residential care facility) or in a non-institutionalized setting where the subject is not living alone and is receiving 24-hour supervision via home health care or a family member. Subjects must have been at their current location for at least 14 days before screening and plan to remain at the same location for the duration of the trial.
* Diagnosis of Dementia (NCD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) Criteria for at least 6 months prior to screening.
* Mini-Mental State Examination (MMSE) < 26.
* Clinically relevant Behavioral and Psychological Symptoms of Dementia (BPSD) operationally defined as NPI-NH agitation/ aggression sub score of ≥3 at screening.
* Documented history of clinically relevant BPSD.
* Ability to participate in study evaluation and ingest oral medication.
* Subjects will be on stable concomitant medications regimen for the treatment of BPSD for at least one month prior to the screening visit.
* Subjects will be on stable concomitant medications regimen for the treatment of concurrent conditions for at least one month prior to the screening visit.

Exclusion Criteria:

* Patients receiving any of the following medications: Astemizole, Cisapride, Pimozide or Terfenadine.
* The agitation/aggression is attributable to concomitant medications, environmental conditions or psychiatric condition.
* Patients with severe heart disease.
* Subjects suffering from Epilepsy.
* Subjects suffering from anxiety disorder.
* Subjects who had psychiatric condition in the past OR suffering from psychosis.
* Schizophrenia OR family history of Schizophrenia OR any other mental disorder.
* Subjects with any other condition, which in the judgment of the investigator would prevent the subject from completing the study.
* Any condition that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the patient.
* Patients suffering from alcohol and/or substance abuse
* Surgery within 30 days prior to screening or scheduled surgery during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-18 (Actual)

PRIMARY OUTCOMES:
Change in score of Cohen-Mansfield Agitation Inventory (CMAI) | week 16
  Proportion of subjects achieving a decrease of four or more points on the Cohen-Mansfield Agitation Inventory (CMAI), a 29-item scale that measures the types and frequencies of agitated behaviors, each rated on a 7-point scale of frequency, where higher scores indicate greater agitation severity.

SECONDARY OUTCOMES:
Change in score of Neuropsychiatric Inventory-Nursing Home Version (NPI-NH) | week 16
  Proportion of subjects with change in score of Neuropsychiatric Inventory-Nursing Home Version (NPI-NH). The greater the NPI-NH score, the more severe and frequent the behavioral disturbances

CONTACTS AND LOCATIONS:
Overall Officials: Vered Hermush, Dr, Principal Investigator — Laniado Hospital Geriatric Department
Locations (1):
- Laniado Hospital, Netanya, Israel

REFERENCES:
- [Derived] Hermush V, Ore L, Stern N, Mizrahi N, Fried M, Krivoshey M, Staghon E, Lederman VE, Bar-Lev Schleider L. Effects of rich cannabidiol oil on behavioral disturbances in patients with dementia: A placebo controlled randomized clinical trial. Front Med (Lausanne). 2022 Sep 6;9:951889. doi: 10.3389/fmed.2022.951889. eCollection 2022. PMID 36148467
- [Derived] Bosnjak Kuharic D, Markovic D, Brkovic T, Jeric Kegalj M, Rubic Z, Vuica Vukasovic A, Jeroncic A, Puljak L. Cannabinoids for the treatment of dementia. Cochrane Database Syst Rev. 2021 Sep 17;9(9):CD012820. doi: 10.1002/14651858.CD012820.pub2. PMID 34532852
- [Derived] Solomon HV, Greenstein AP, DeLisi LE. Cannabis Use in Older Adults: A Perspective. Harv Rev Psychiatry. 2021 May-Jun 01;29(3):225-233. doi: 10.1097/HRP.0000000000000289. PMID 33660625